CLINICAL TRIAL: NCT06927622
Title: Study on the Influence of Corona Virus Disease 2019 on Obstetric Outcome and Offspring Development
Brief Title: Corona Virus Disease 2019 Cohort Study
Status: Recruiting | Type: Observational
Sponsor: Shandong University (Other)
Collaborators: Qilu Hospital of Shandong University (Other); Jinan Maternity and Child Health Care Hospital (Unknown); Shandong Provincial Maternity and Child Health Care Hospital (Unknown); The Second Hospital of Shandong University (Other); Qianfoshan Hospital (Other)
Responsible Party: Principal Investigator, Yinuo Song, Principal Investigator, Shandong University
Other Study IDs: LL202303018
Record Dates: First submitted 2023-11-27; First posted 2025-04-15 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: COVID-19 Pneumonia; COVID-19 Pandemic; COVID-19
Keywords: pregnant woman; birth cohort; infant; nervous system development
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The goal of this observational study is to learn about the influence of Corona Virus Disease 2019 on obstetric outcome and offspring development.

DETAILED DESCRIPTION:
The main questions it aims to answer are:

* Collect the information about Corona Virus Disease 2019 infection and medication of pregnant women to establish a birth cohort, and analyze the correlation between Corona Virus Disease 2019 infection during pregnancy and adverse pregnancy outcomes and birth outcomes.
* The offspring born in this cohort were followed up to analyze the effects of Corona Virus Disease 2019 infection during pregnancy on the nervous system development of the offspring.

Researchers will compare Corona Virus Disease 2019 infection group and uninfected group during pregnancy to see if Corona Virus Disease 2019 infection has adverse effects on pregnant women and their offspring.

ELIGIBILITY:
Inclusion Criteria:

* Conduct regular prenatal examinations in the hospital and establish a pregnancy and childbirth health manual, planning for pregnant women who are hospitalized for delivery;
* Conduct regular physical examinations in the hospital and establish a children's health manual for infants.
* Age ≥ 18 years old

Exclusion Criteria:

* Concomitant tumor related diseases;
* Individuals with severe mental disorders.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The population of this study is pregnant women who undergo regular prenatal examinations in hospitals, establish a prenatal care manual, plan hospital delivery, have no comorbid tumor diseases, are mentally normal, and are aged ≥ 18 years old.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Measure the developmental outcomes of the nervous system using the Gesell Development Plan (GDS) or the 0-6-year-old Child Development Scale (DST). | From 6 months of birth to completion of the GDS measurement, the assessment is up to 6 months
  GDS mainly diagnoses four abilities: motor ability, object ability, speech ability, and human ability,. Thus, the development quotient of four aspects can be obtained. If the development quotient is below 65-75, it indicates serious backwardness. The DST assessment includes five functional areas: gross motor, fine motor, language, adaptability, and social behavior, to obtain developmental quotient, which is used to measure the developmental behavior of children and evaluate their level of development. A score above 130 indicates excellent performance, and a score below 70 indicates intellectual development disorder.
Pregnancy complications or comorbidities | Starting prenatal examination until discharge，the evaluation take up to 10 months
  Obtain relevant information from medical records. Pregnancy complications refer to non pregnancy related diseases that occur before or during pregnancy, while pregnancy complications refer to any diseases that coexist with pregnancy.
Obtain neonatal outcomes. | The evaluation period from birth to discharge is up to 1 week
  Obtain neonatal outcomes from neonatal records, including macrosomia, neonatal asphyxia, fetal distress, low birth weight infants, and deformed infants.
Comprehensive results of COVID-19 infection during pregnancy | Baseline data were obtained when participants were enrolled in the study and assessed for up to 1 years
  Through questionnaires, medical records and test sheets, The investigators can get whether the pregnant women have been infected with COVID-19 during pregnancy, the time of infection, pregnancy weeks, symptoms, etc.

SECONDARY OUTCOMES:
Delivery method | The evaluation period from admission to delivery to discharge is up to 1 week
  Natural delivery, vaginal surgery, or curettage.
Estimation of bleeding volume | The evaluation period from admission to delivery to discharge is up to 1 week
  Total amount of bleeding during or 24 hours postpartum.

CONTACTS AND LOCATIONS:
Overall Officials: Fanzhen Hong, Doctorate, Study Director — The Second Hospital of Shandong University; Xia Luo, Doctorate, Study Director — Qilu Hospital of Shandong University; Yueqin Xu, Doctorate, Study Director — Qianfoshan Hospital; Qiuhong Yang, Doctorate, Study Director — Jinan Maternity and Child Health Care Hospital; Jie Chen, Doctorate, Study Chair — Shandong University; Yinuo Song, Master, Principal Investigator — Shandong University
Locations (5):
- China (5):
  - The Second Hospital of Shandong University, Jinan, Shandong
  - Jinan Maternity and Child Health Care Hospital, Jinan
  - Qianfoshan Hospital, Jinan
  - Qilu Hospital of Shandong University, Jinan
  - Shandong Provincial Maternity and Child Health Care Hospital, Jinan

IPD SHARING:
Plan to Share IPD: Yes
The investigators will only allow users to use the data and supporting files based on a clear data sharing agreement, which enforces (a) their commitment to use the data only for research purposes and will not identify any individual study participants; (b) Promise to use appropriate technology to protect all research data; (c) Prohibit the redistribution of data to third parties and appropriately confirm data resources, as well as (d) commit to destroying and/or returning data after analysis is completed. Co investigators can access data collected as part of their purpose. The investigators involved in this project can only access the data through the chief investigator. The investigators will regularly monitor data to maintain security, safety, and productivity.
Supporting Information: Study Protocol
Time Frame: The investigators will be provided within 1 Year after the release of the main research findings
Access Criteria: Access is only provided after submitting research proposals and obtaining approval from an independent review team, as well as after the data sharing agreement is in place.